CLINICAL TRIAL: NCT04535869
Title: Efficacy and Safety of Direct Anti HCV Drugs in the Treatment of SARS-COV-2 (COVID-19)
Acronym: CCOVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Elbendary, Professor of Tropical Medicine and Hepatogastroenterology, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.20.08.1214
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: COVID; Anti- HCV drugs,; Sofosbuvir; Daclatasvir; DAAs; Efficacy
MeSH Terms: conditions — COVID-19 | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A)standard therapy group (No Intervention): No intervention COVID- 19 patients who received a standard therapy group according to the ministry of health protocol
- B)Standard Therapy group plus Ant-HCV drugs (Active Comparator): Intervention COVID- 19 patients who received a standard therapy group according to the ministry of health protocol plus sofosbuvir 400 mg and Daclatasvir 200mg
  Interventions: Drug: Sofosbuvir 400 MG plus Daclatasvir 200mg

INTERVENTIONS:
Drug: Sofosbuvir 400 MG plus Daclatasvir 200mg — This group which receive sofosbuvir and daclatasvir for 14 days plus standard therapy
  Other Names: Direct antiviarl agents
  Arms: B)Standard Therapy group plus Ant-HCV drugs

SUMMARY:
COVID 19 which started from a zoonotic transmission related to crowded markets was confirmed to have a high potential for transmission to close contacts on 20 January 2020 by the National Health Commission of China and it was announced as a pandemic by the WHO on 11 March 2020.

There is currently no clinically proven specific antiviral agent available for SARS-CoV-2 infection. Supportive treatment, including oxygen therapy, conservation fluid management, and broad-spectrum antibiotics to cover secondary bacterial infection, remains the most important management strategy.

Interestingly, sofosbuvir has recently been proposed as an antiviral for the SARS-CoV-2 based on the similarity between the replication mechanisms of the HCV and the coronaviruses.

Aim of our study is to assess the safety and efficacy of of the addition of HCV treatment to the standard regimen for the treatment of patients according to MOHP protocol.

DETAILED DESCRIPTION:
SARS-CoV-2 infection have a wide clinical spectrum ranging between asymptomatic infection, mild upper respiratory tract symptoms, and severe viral pneumonia (fever, malaise, dry cough, shortness of breath, and respiratory distress) that may result in respiratory failure and finally death.

There is currently no clinically proven specific antiviral agent available for SARS-CoV-2 infection. Supportive treatment, including oxygen therapy, conservation fluid management, and broad-spectrum antibiotics to cover secondary bacterial infection, remains the most important management strategy.

For direct antiviral treatment of SARS-CoV-2, the China International Exchange and Promotive Association for Medical and Health Care (CPAM) recommended usage of lopinavir; ritonavir. Their recommendation was based on weak evidence from retrospective cohort, historically controlled studies, case reports, and case series reporting a clinical benefit of lopinavir; ritonavir in the management of other coronavirus infection [i.e., SARS-CoV 1 and Middle East respiratory syndrome coronavirus (MERS-CoV)] .

However, the first randomized clinical trial with lopinavir/ritonavir demonstrated no benefit over standard care in 199 hospitalized adults with severe COVID-19. There is no evidence to support the use of other antiretrovirals, including protease inhibitors; indeed, structural analysis demonstrates no darunavir binding to COVID-19 protease A group of Korean physicians experienced in SARS-CoV-2 infected patients' treatment developed recommendations for the treatment of COVID-19. According to them, antiviral medications lopinavir 400 mg; ritonavir 100 mg, or chloroquine is considered to be used in older patients or patients with chronic health conditions and life-threatening symptoms. If chloroquine is unavailable, hydroxychloroquine is recommended. Both of them have reported the ability of inhibition of SARS-CoV-2 in vitro.

CPAM guidelines included them as they were associated with reduced progression of the disease and decreased duration of symptoms. In an open-label study of 36 patients with COVID-19, the use of hydroxychloroquine (200 mg three times per day for 10 days) was associated with a higher rate of undetectable SARS-CoV-2 RNA on nasopharyngeal specimens at day 6 compared with no specific treatment (70 versus 12.5 percent). In this study, the use of azithromycin in combination with hydroxychloroquine appeared to have an additional benefit, but there are methodologic concerns about the control groups for the study, and the biologic basis for using azithromycin in this setting is unclear. In the United States, the FDA issued an emergency use authorization to allow the use of these agents in adolescents or adults hospitalized for COVID-19.

One of the studies done on SARS-COV-1 strongly suggested that using ribavirin as therapy should be reconsidered until further animal studies clarify the effects of ribavirin on cytokine and chemokine profiles during infection and until ribavirin can be demonstrated to have a significant effect on reducing viral replication in vivo. Data from a molecular docking experiment using the SARS-CoV-2 RNA dependent RNA polymerase (RdRp) model identified the tight binding of sofosbuvir and ribavirin to the coronavirus RdRp, thereby suggesting possible efficacy of sofosbuvir and ribavirin in treating the COVID-19 infection.

A three-dimensional model of the SARS-CoV-2 (aka 2019-nCoV) 3C-like protease (3CL ) was prepared then performed virtual screening for purchasable drugs checking the actions, targets, and side effects of the 16 candidates. Velpatasvir and ledipasvir are examples of these drugs ( which are inhibitors of the NS5A protein of the hepatitis C virus (HCV). Both are marketed as approved drugs in combination with sofosbuvir, which is a prodrug nucleotide analog inhibitor of RNA-dependent RNA polymerase (RdRp, or NS5B).

Interestingly, sofosbuvir has recently been proposed as an antiviral for the SARS-CoV-2 based on the similarity between the replication mechanisms of the HCV and the coronaviruses.

Based on this data it was suggested that these dual-component HCV drugs, Epclusa (velpatasvir/sofosbuvir) and Harvoni (ledipasvir/sofosbuvir), may be attractive candidates to repurpose because they may inhibit two coronaviral enzymes. A drug that can target two viral proteins substantially reduces the ability of the virus to develop resistance. These direct-acting antiviral drugs are also associated with very minimal side effects and are conveniently orally administered.

The aim of this study is to assess the safety and efficacy of the addition of HCV treatment to the standard regimen for the treatment of COVID-19 patients according to MOHP protocol .

ELIGIBILITY:
Inclusion Criteria:

* All cases positive for COVID-19
* Male and non-pregnant female patients,
* 18 years of age or older,
* All moderate and severe caseswith pneuomnia.

Exclusion Criteria:

* Known allergy or hypersensitivity to the used medications
* Known severe liver disease
* Use of medications that are contraindicated with the trial medications and that could not be replaced or stopped during the trial period
* Pregnancy or breast-feeding or known active HCV infection, because of concerns about the development of resistance
* History of bone marrow transplant
* Known G6PD deficiency
* Chronic hemodialysis or Glomerular Filtration Rate < 20ml/min
* Psoriasis
* Porphyria
* Concomitant use of digitalis, flecainide, amiodarone, procainamide, or propafenone
* Known history of long QT syndrome
* Current known QTc>500 msec
* Pregnant or nursing
* Weight < 35kg
* Seizure disorder
* Patients receiving Amiodarone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-09-03 (Estimated)

PRIMARY OUTCOMES:
rate of virological cure by Rt -PCR for COVID -19using the triple therapy as compared to standard treatment | for every case must be done after 2 weeks from the start of treatment.
  All PCR for COVID must be negative

SECONDARY OUTCOMES:
resolution of pneumonia BY high resolution Computed tomography | Computed tomography must be done after 2 weeks to detect resolution of pneumonia
  clinical status as assessed by earlier resolution of pneumonia in the intervention arm when compared to the control group

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Faculty of Medicine, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hallin RW. Femoropopliteal versus femorotibial bypass grafting for lower extremity revascularization. Am Surg. 1976 Jul;42(7):522-6. PMID 937862
- [Background] Depo-Provera may be linked to uterine cancer, preliminary data imply. Fam Plann Perspect. 1979 Jan-Feb;11(1):47. No abstract available. PMID 105932
- [Background] O'Brien PJ, Hawco FJ. Hydroxyl-radical formation during prostaglandin formation catalysed by prostaglandin cyclo-oxygenase [proceedings]. Biochem Soc Trans. 1978;6(6):1169-71. doi: 10.1042/bst0061169. No abstract available. PMID 105949
- [Background] Kirkegaard C, Faber J, Hummer L, Rogowski P. Increased levels of TRH in cerebrospinal fluid from patients with endogenous depression. Psychoneuroendocrinology. 1979 Jul;4(3):227-35. doi: 10.1016/0306-4530(79)90006-4. No abstract available. PMID 117477
- [Result] Phelan AL, Katz R, Gostin LO. The Novel Coronavirus Originating in Wuhan, China: Challenges for Global Health Governance. JAMA. 2020 Feb 25;323(8):709-710. doi: 10.1001/jama.2020.1097. No abstract available. PMID 31999307